

UNICANCE PAYS DE LA LOIRE

Short Title: APA Ref ICO: ICO-2020-05 ID-RCB: 2020-A00275-34

**SYNOPSIS** 

| | ADA |
|---|---|
| SHORT TITLE / OFFICIAL TITLE | APA Prospective Evaluation of the Impact on Patients' Quality of Life of a 12-Week Adapted Physical Activity Program (APA) at Institut de Cancerologie de l'Ouest (ICO) |
| SPONSOR | Institut de Cancerologie de l'Ouest (ICO) |
| INVESTIGATOR COORDINATOR | Dr Sophie ABADIE-LACOURTOISIE Oncologue Médical |
| METHODOLOGIST / STATISTICIAN | Dr Valérie SEEGERS And Catherine GUERIN-CHARBONNEL Institut de Cancérologie de l'Ouest Direction de la Recherche Clinique (DRC) |
| OBJECTIVES | Primary: Describe the changes in quality of life experienced by cancer patients treated at the ICO site in Angers who participated in the ICO's 12-week adapted physical activity program. Secondary: a) Describe attendance at the APA program. b) Measure changes in kinesiophobia. c) Measure physical activity at the start of the APA program. |
| METHODOLOGY | This is a prospective, non-comparative, monocenter cohort study with the administration of a quality-of-life questionnaire. |
| TARGET POPULATION | Adult subjects enrolled in the APA program at ICO (Angers site) during the first semester of 2020, regardless of cancer type and ongoing treatment (chemotherapy, radiotherapy, hormone therapy, immunotherapy). |
| NUMBER OF PATIENTS | All patients meeting the eligibility criteria. About 70 patients. |
| NUMBER OF CENTRES | 1 – ICO Site Angers |
| STATISTICAL ANALYSIS | This is a descriptive study aiming to characterize the quality of life of cancer patients during their APA program. A flowchart will be created to define the completion rate of questionnaires at different time points. Baseline characteristics of the population will be described. Quantitative data will be summarized using mean, standard deviation, median, minimum, maximum, and 25th and 75th percentiles. Categorical or binary data will be summarized by distribution across categories and expressed as percentages. The number of missing data will be reported. No imputation procedure for missing data is planned. Individual trajectories of FACIT scores will be graphically presented with sample sizes clearly indicated at each time point. Scores (quantitative data) will be summarized at the three measurement times. A paired data comparison will be performed to compare scores across time points. TAMPA scores (quantitative data) will be graphically presented using boxplots. |